CLINICAL TRIAL: NCT05824364
Title: Exercise aNd hEArt Transplant
Acronym: ENEA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Don Carlo Gnocchi Onlus (Other)
Responsible Party: Principal Investigator, Nuccia Morici, Head of Cardiac Rehabilitation Department, Fondazione Don Carlo Gnocchi Onlus
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ENEA
Record Dates: First submitted 2023-01-16; First posted 2023-04-21 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Heart Transplant
Keywords: cardiac rehabilitation; telerehabilitation; rehabilomics
MeSH Terms: interventions — Telerehabilitation

STUDY DESIGN:
Intervention Model Description: parallel and cross over designs will be adopted according to the specific purposes of that given clinical study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Case (Experimental): two-four weeks of on-site cardiac rehabilitation (CR) followed by 12 weeks of telerehabilitation
  Interventions: Other: telerehabilitation; Other: rehabilomic
- Control (Active Comparator): 4 weeks of on-site standard CR
  Interventions: Other: rehabilomic

INTERVENTIONS:
Other: telerehabilitation — Telerehabilitation activites will be tested with the aim to provide 1) continuation of rehabilitative care, focused on physical training and patients'monitoring , and 2) information in the mid-term about study goals.
  Arms: Case
Other: rehabilomic — blood withdrawal (10 ml of blood, two tubes of 5 ml for serum isolation): at the hospital admission at the Cardiac Rehabilitation Unit of IRCCS Fondazione Don Gnocchi of Milan (T0) and after the rehabilitative treatment (T1)

SUMMARY:
Registry-based randomized clinical trial (RRCT) to assess the safety and efficacy of two different schemes of exercise training in patients who have recently undergone heart transplantation

DETAILED DESCRIPTION:
40 patients who achieved Heart transplantation (HTx) will be randomized in a pilot study to 4 weeks of on-site standard CR (control arm) versus two-four weeks of on-site CR followed by 12 weeks of telerehabilitation (experimental arm). Both surrogate endpoints [cardiometabolic equivalents (Vo2 peak)] and clinical endpoint [primary outcome defined as acute rejection, hospitalization for heart failure, stroke, myocardial infarction, all-cause mortality, at the longest follow-up available (minimum 6-month follow-up)] will be evaluated.

The rehabilomic approach will be applied in order to identify specific patients' phenotype. To identify the potential variations of circulating molecules levels that could be indicators of the rehabilitation outcome and/or progression of the disease, the research team will focus on the analysis of extracellular vesicles (EVs) isolated from the serum of the 40 patients at admission (T0) and after cardiac rehabilitation (T1). In particular, researchers will detect and analyze the relative amount of serum EVs derived from platelets, endothelium, cardiomyocytes, and macrophages, as their levels are reported to be associated with the occurrence of heart failure.

ELIGIBILITY:
Inclusion Criteria:

* All the patients admitted in the on-site CR after HTx

Exclusion Criteria:

* unable to sign informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-05-20 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-11-28 (Estimated)

PRIMARY OUTCOMES:
Cardiovascular events | 6-months
  Incidence of acute rejection, Rate of hospitalization for heart failure, Incidence of stroke, Incidence of myocardial infarction and incidence of all-cause mortality

SECONDARY OUTCOMES:
Vo2 peak | 6-months
  cardiometabolic equivalents (Vo2 peak)
extracellular vesicles (EVs) analysis with Surface Plasmon Resonance imaging (SPRi) | up to 4 weeks
  EVs will be isolated from blood, characterized by standard procedures and injected on the SPRi biosensor for the differential quantification of multiple EV subfamilies. The expression of a secondary antigen will be evaluated on the surface of immobilized EVs.
EuroQol 5-Dimension (EQ-5D-5L) | 6-months
  The EQ-5D-5L is a generic questionnaire measuring five domains of current health-related quality of life, where a higher index score indicates higher health-related quality of life.
Short Form 36 (SF36) | 6-months
  The 36-Item Short Form Health Survey (SF-36) is a set of generic, coherent, and easily administered quality-of-life measures.
Hospital Anxiety and Depression Scale (HADS) | 6-months
  The HADS is a 14-item generic questionnaire measuring symptoms of anxiety and depression within the last week.

CONTACTS AND LOCATIONS:
Overall Officials: Nuccia Morici, MD, Principal Investigator — IRCCS Fondazione Don Carlo Gnocchi, Milan, Italy
Locations (1):
- IRCCS Fondazione Don Gnocchi, Milan, Milan, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pedersini P, Picciolini S, Di Salvo F, Toccafondi A, Novembre G, Gualerzi A, Cusmano I, Garascia A, Tavanelli M, Verde A, Masciocco G, Ricci C, Mannini A, Bedoni M, Morici N. The Exercise aNd hEArt transplant (ENEA) trial - a registry-based randomized controlled trial evaluating the safety and efficacy of cardiac telerehabilitation after heart transplant. Contemp Clin Trials. 2024 Jan;136:107415. doi: 10.1016/j.cct.2023.107415. Epub 2023 Dec 17. PMID 38114046